CLINICAL TRIAL: NCT06676787
Title: Demand Side Incentives Project (DSI)
Brief Title: Evaluating the Impact of Demand-Side Incentives (DSI) on Zero Dose Burden and Immunisation Coverage in Nigeria
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Corona Management Systems (Other)
Collaborators: Kwara State Primary Healthcare Development Agency (Unknown); Oyo State Primary Healthcare Board (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NHREC/01/01/2007-13/09/2023
Record Dates: First submitted 2024-10-21; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Incentives
Keywords: Nigeria; Immunisation; Incentives; Caregivers

STUDY DESIGN:
Intervention Model Description: The interventions for each arm were selected based on findings from a feasibility evaluation conducted with national and sub-national stakeholders. This evaluation considered the local context of immunisation challenges and identified incentives that have broad stakeholder support across the Expanded Programme on Immunization (EPI) and the community.
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (Experimental): Wards in Kwara and Oyo states, where the DSI project provides transportation vouchers to children after vaccination, provided they are aged 0-23 months and reside in communities within the ward.
  Interventions: Other: Transportation Voucher, Comunity engagement and microplannnig support
- Arm 2 (Experimental): Wards in Kwara and Oyo states, where the DSI project provides monthly financing to routine immunisation primary healthcare facilities to support immunisation and other health services, provided these health facilities are located within the ward.
  Interventions: Other: Direct Facility Funding, Community Engagement, and Microplaning Support
- Arm 3 (Experimental): Wards in Kwara and Oyo states, where the DSI project provides transportation vouchers to children after vaccination, provided they are aged 0-23 months and reside in communities within the ward and also provides monthly financing to routine immunisation primary healthcare facilities to support immunisation and other health services, provided these health facilities are located within these wards.
  Interventions: Other: Transportation Voucher, Direct Facility Funding, Community engagement and Microplanning support
- Control (No Intervention): No intervention in these wards

INTERVENTIONS:
Other: Transportation Voucher, Comunity engagement and microplannnig support — Transportation vouchers will be provided to caregivers of eligible children after vaccination at designated routine immunisation health facilities. This is in addition to support for microplaning (technical assistance) for these routine immunisation health facilities and comunity engagement at their catchment areas.
  Arms: Arm 1
Other: Direct Facility Funding, Community Engagement, and Microplaning Support — Direct funding will be provided to designated routine immunisation health facilities monthly, in addition to weekly performance monitoring and quarterly financial capacity building. Also, there will be support for microplaning (technical assistance) for these routine immunisation health facilities and comunity engagement at their catchment areas.
  Arms: Arm 2
Other: Transportation Voucher, Direct Facility Funding, Community engagement and Microplanning support — Transportation vouchers will be provided to caregivers of eligible children after vaccination at designated routine immunisation health facilities. Direct funding will be provided to designated routine immunisation health facilities monthly, in addition to weekly oerformance monitoring and quarterly financial capacity building. Also, there will be support for microplaning (technical assistance) for these routine immunisation health facilities and comunity engagement at their catchment areas.
  Arms: Arm 3

SUMMARY:
The goal of this cluster Randomised Controlled Trial (cRCT) is to evaluate the impact and effectiveness of demand-side incentives (DSIs) in improving immunisation coverage and reducing the burden of zero-dose children between the age of 12-23months in Nigeria.

The study seeks to answer the following questions

1. What is the impact of demand-side incentives on increasing immunization coverage in the selected subnational regions of Nigeria?
2. What is the effect of demand-side incentives on reducing the zero-dose burden in selected subnational regions in Nigeria?
3. What is the effect of various demand-side incentive schemes on improving the timeliness of vaccination among children aged 0 to 23 months in the selected subnational regions of Nigeria?
4. What is the impact of different demand-side incentive schemes on enhancing the immunization knowledge and perception of caregivers with children aged 0 to 23 months in the selected subnational regions Nigeria by December 2025.

DETAILED DESCRIPTION:
Background Immunisation coverage is a critical aspect of public health, as it protects children from vaccine-preventable diseases and deaths. However, according to World Health Organisations and United Nations Children's Education Fund, WHO/UNICEF Estimates of National Immunisation Coverage (WUENIC) data, approximately 25 million children worldwide missed out on life-saving vaccines in 2021, an increase of 6 million compared to 2019. This included 18.2 million zero-dose children, with more than 60% of them living in ten countries, including Nigeria. The global coverage of the third dose of diphtheria-tetanus-pertussis (DTP3) also declined from 86% in 2019 to 81% in 2021 according to the same WUENIC reports, the lowest level since 2008. Several factors have been identified as potentially contributing to this decline, such as increased conflict and fragile settings, misinformation, and disruptions caused by the Corona Virus Disease 2019 (COVID-19) pandemic, including service and supply chain disruptions and resource diversion to pandemic response efforts. The 2022 WUENIC results however show that vaccination coverage has started to improve following on from the decline in the preceding years.

Each year, nearly 2.5 million children living in Nigeria do not receive DTP1, and in 2020, an additional 500,000 children were unvaccinated because of the COVID-19 pandemic. In Nigeria, DTP1 coverage was reported in the 2022 Multiple Indicator Cluster Survey (MICS) to be 68%. The 2021 WHO/UNICEF estimates of national immunisation coverage (WUENIC) report a DTP1 coverage of 70%. Data from the District Health Information System 2 (DHIS 2) for 2022 shows cumulative DTP1 national coverage at 90.95%. These differences in coverage contribute to the challenges of visibility into where and why zero dose children exist.

The Equity Reference Group for Immunisation (ERG) has emphasised and called for a greater focus on four key areas to reach Zero dose children, namely conflict-affected, urban poor, and remote rural areas as well as gender-related barriers. Factors that have been reported to drive the existence of zero dose children in Nigeria include maternal education, fears and misconceptions, and access to health facilities, many of which are intricately linked to the four key areas identified by the ERG. Approximately 55% of zero-dose children in Nigeria however are concentrated in seven states - Kano, Sokoto, Bauchi, Katsina, Niger, Zamfara and Kaduna and are at greater risk of becoming sick or dying from preventable diseases. Sub-national variations in coverage exist, with Lagos and Kano states contributing the largest burden of zero-dose children despite significant differences between the state level coverages.

Inequities in immunisation coverage are reportedly common in urban areas affecting the urban poor, who often live in urban slums. Cumulative DTP1 coverages higher than 100% are unfortunately not uncommon on the DHIS 2, appearing to be reported more often among urban LGAs than among rural LGAs. In-country stakeholders largely attribute this data quality issue to the denominator used to calculate the coverage, as this denominator is based on the projected growth rates from the 2006 population census. The factors around geographical location however run deeper than the level of the LGA with administrative data on the DHIS 2 also showing disparities in DTP1 coverage between health facilities. Nigeria also has communities that have or are still experiencing conflicts, contributing to limited access to immunisation services in these communities and increased number of zero-dose children.

To improve immunisation coverage, Nigeria adopted the Reach Every Ward (REW) strategy in 2005, the REW strategy focuses on routine immunisation in health facilities and outreaches, including components such as improved access for under-served and hard-to-reach areas; supportive supervision; monitoring and use of data for action; community mobilisation and improving community links with service delivery. The National Emergency RI Coordination Centre (NERICC) implements the Optimised Integrated Routine Immunisation Sessions (OIRIS) approach with five key pillars: optimised Routine Immunisation (RI) sessions, integration with other services, intensified supportive supervision, ownership, and accountability. OIRIS aims to enhance RI service access by removing barriers through improved microplan development and implementation in states and Local Government Areas (LGAs). OIRIS also drives the implementation of the revised community engagement strategy, with community level line-listing of newborns to support connection to immunisation services, as a complement to other communications and demand generation activities and strategies.

Gavi, in partnership with Corona Management Systems, has launched an innovative Demand-Side Incentive (DSI) Programme to strengthen immunisation programmes in Cameroon, the Democratic Republic of Congo, Lesotho, and Nigeria. The programme aims to increase vaccination coverage, reach marginalised communities, improve timeliness, and enhance caregivers' attitudes towards vaccination.

Rationale Globally, approximately two-thirds of Zero-dose children live in households that survive on less than US$ 1.90 per day and it is estimated that over 11% of Zero-dose children are living in remote,-rural areas, 26% in urban and peri-urban areas, and between 6 and 18% in conflict-affected locations. The Equity Reference Group for Immunisation (ERG) has emphasised and called for a greater focus on four key areas to reach Zero-dose children, namely conflict-affected, urban poor, and remote rural areas as well as gender-related barriers. The Gavi 5.0 strategy prioritises 'Leaving no one behind with immunisation', yet gaps are still in knowledge on many of the structural determinants of zero-dose, and on where and why zero-dose children and missed communities are still a challenge.

The Gavi 5.0 Strategy (2021-2025) recognises the need to strengthen health systems to increase equity in immunisation. While Gavi historically focused on supply-side incentives, the strategy also emphasises demand-side initiatives (DSI). DSI have shown promising outcomes in improving the demand and coverage of health services, including vaccination. DSI have been implemented in various low- and middle-income countries, including Nigeria with positive results. These initiatives often combine cash and non-cash incentives to drive health-seeking behaviours. It is important to consider the cost of fully vaccinating a child, which is estimated to be between US$25 and $45, excluding non-vaccine costs such as service delivery, training, supervision, monitoring, and demand generation. While governments have made progress in increasing funding for immunisation programmes, further commitment is needed to achieve full financing and national ownership of these programmes. DSI have proven value as an innovative instrument to help address the challenge of zero-dose and missed communities. There is however an ardent desire that the DSI are low-cost, providing a pathway for future transitioning to country governments and for sustainability.

There is also a broad recognition of the importance of implementing DSI across different segments of Gavi priority countries. This would potentially provide a platform to show alignment with current approaches and other interventions of the alliance. In this regard, Nigeria would fall into the category of high-impact countries, with pockets of conflict. As part of the country selection process, particular attention has been paid to countries with low DTP-1 national coverage. Nigeria faces significant challenges in immunisation coverage. Nigeria has over 2 million zero-dose children, contributing significantly to the global burden of under-immunised children. There are also differences in the burden of zero-dose children in sub-national geographies due to differences in population and immunisation coverages. The DTP3 national coverage in Nigeria is 56%, showing a substantial number of children who are not receiving the recommended vaccinations.

In selecting Nigeria for the DSI project, factors such as the absolute population of zero-dose children, sub-national variations, equity considerations (such as urban poor and rural hard-to-reach populations), conflict and fragile settings, and gender-related barriers were considered. The choice also considered the countries' historical experiences with implementing DSI and the appetite for such interventions. The Investigators find this important as it helps corroborate country appetite for DSI in the past and helps provide a platform of key lessons of what has worked and what did not work within the specific country context. Country appetite for implementing DSI was also set up from our preliminary engagements with Expanded Programme on Immunisation (EPI) stakeholders, as another fundamental driver. This will ultimately define appetite for collaboration and can make or mar successful implementation. In Nigeria, New Incentives provide Conditional Cash Transfers (CCT) to caregivers who complete the full schedule of routine immunisation for their children. Also in Nigeria, the Subsidy Reinvestment and Empowerment Programme (SURE-P) which invested profits from fuel revenues into a social protection fund for vulnerable populations disbursed cash transfers upon completion of routine immunisation.

Country presence of the implementing team and earlier work experiences in select countries and local understanding of cost of living and human development indices, were also key parameters that shaped our choice. These were very instrumental to stakeholder management and will provide a pathway to identifying, selecting, and engaging with local partners. Corona Management Systems has the country presence and a history of implementing projects collaboratively in Nigeria. Corona Management Systems also has a strong understanding on co-creating the DSI project with the National Primary Healthcare Development Agency and partners, to ensure that the project design is robust, fit for purpose for the country, and complements other ongoing interventions and investments.

In summary, Nigeria has low national immunisation coverage, substantial burden of zero-dose children, previous experience with DSI, and the country's appetite for implementing DSI makes it an ideal candidate for this project. The Demand-Side Incentives (DSI) to Address Immunisation Challenges project will therefore be implemented in four countries: Cameroon, Democratic Republic of Congo (DRC), Lesotho, and Nigeria. In Nigeria, Oyo and Kwara states have been selected for the implementation of the DSI project. The project Implementation will utilise an experimental design. The unit of experimentation will be the sub-district level, and each unit will constitute a cluster. In Nigeria, this sub-district level will be at the level of the political ward.

OBJECTIVES OF THE STUDY

The objective of this cluster Randomised Controlled Trial (cRCT) is to evaluate the impact and effectiveness of demand-side incentives (DSI) in improving immunisation coverage and reducing the burden of zero-dose children in Nigeria. The study aligns with the Immunisation Agenda 2030, the Gavi 5.0 strategy, and the country's priorities in strengthening the immunisation programme. The specific objectives of this cRCT include:

* Assess the impact of demand-side incentives on increasing immunization coverage in the selected subnational regions of Nigeria, by December 2025.
* Assess the effect of demand-side incentives on reducing the zero-dose burden in selected subnational regions in Nigeria, by December 2025.
* Examine the effects of various demand-side incentive schemes on improving the timeliness of vaccination among children aged 0 to 23 months in the selected subnational regions of Nigeria, by December 2025.
* Explore the impact of different demand-side incentive schemes on enhancing the immunization knowledge and perception of caregivers with children aged 0 to 23 months in the selected subnational regions Nigeria by December 2025.

SCOPE OF THE STUDY Thematic Scope

The cluster Randomised Controlled Trial (cRCT) aims to evaluate the impact and effectiveness of demand-side incentives (DSI) in improving immunisation coverage and reducing the burden of zero-dose children in Nigeria. Key areas of focus for the study include:

1. A review of existing demand-side incentives and their impact on immunisation coverage and equity.
2. Behavioural and social drivers of vaccination uptake and vaccination service utilisation by the target population.
3. Structural determinants of zero-dose children in different settings (e.g., distant rural areas, urban poor settings, conflict-affected regions, areas with gender-related barriers).
4. Identification of primary challenges and opportunities through a baseline evaluation to inform the design and implementation of the Demand-Side Incentive (DSI) Programme to strengthen immunisation programmes; and
5. Evaluation of the impact of demand-side incentives on vaccination coverage, reduction of zero-dose children, improvement of vaccination service timeliness and shifts in behavioural and social drivers of vaccination uptake.

Geographic Scope The study will be conducted in selected Oyo and Kwara State in Nigeria. These areas were identified during the feasibility assessment based on the following criteria: low vaccination (low Penta 3 coverage rate), high burden of zero-dose children (low Penta 1 coverage rate or absolute number of zero-dose children), the absence of any current demand-side incentives intervention, and sustained stakeholder buy-in. The study will specifically target poor and underserved communities, including those in remote and hard-to-reach areas.

Chronological Scope The study will run from August 2024 till December 2025 and will enrol children eligible for routine immunisation in the intervention locations.

METHODOLOGY Study Type This study will employ a pragmatic, parallel cluster Randomised Controlled Trial (cRCT) design to evaluate the impact of the Demand-Side Incentives (DSI) on zero-dose burden and immunisation coverage in intervention LGAs in Nigeria. A pragmatic, parallel cRCT design is a type of research design that aims to evaluate the effectiveness of an intervention in real-world settings, providing insights into how the intervention works in routine practice.

Study Design The study will employ a cRCT design, focusing on the smallest administrative unit in Nigeria, known as a "political ward" or "ward," each with an estimated population of 10,000. These wards will serve as the sub-district level for the study, with each selected ward considered a cluster. The study is structured as a four-arm cRCT, with a total of 480 clusters (120 per arm). These clusters will be randomly divided into four groups: three intervention arms (360 clusters) and one control arm (120 clusters).

Enrolment will occur at the cluster level, meaning all children aged 0-23 months living in a selected cluster will be allocated to the same arm as the cluster. The study will be implemented across an estimated 49 Local Government Areas (LGAs), each typically including an average of ten wards, in selected sub geographies of Nigeria.

The study locations have been chosen for their low immunisation coverage, thereby focusing on areas with a high number of children receiving zero doses of essential vaccines. The sample size has been calculated to enable impact analysis on Zero Dose in these regions.

The interventions for each arm were selected based on findings from a feasibility evaluation conducted with national and sub-national stakeholders. This evaluation considered the local context of immunisation challenges and identified incentives that have broad stakeholder support across the Expanded Programme on Immunization (EPI) and the community.

Study Area and Population The study will be conducted in selected wards within identified Local Government Areas (LGAs) in Oyo and Kwara states of Nigeria. These areas have been chosen due to their immunisation coverage challenges and low performance indicators. The target population for this study will include key stakeholders involved in designing and executing immunisation programme strategies, community-level participants, and caregivers of infants aged 0 to 23 months.

Sampling Strategy

To ascertain the optimal sample size for each cluster (ward) to detect a 15% effect size, the WebPower package was employed within the R programming language. This package facilitated the computation of statistical power analysis for Cluster Randomized Trials (cRCT) with two arms-specifically, comparing the control arm against each implementation arm. The calculation considered the specified effect size, the number of subjects per cluster, intra-class correlation, significance level, and power.

Using an Intra-Class Correlation (ICC) of 0.16, based on relevant literature, and adopting a 95% confidence level, various sample sizes were stimulate. The results depicted revealed that over 80% power could be achieved with sample sizes ranging from 100 to 400. Considering practical implementation feasibility, a sample size of 100 was opted for with 20% margin in case of drop out, making it 120.

ELIGIBILITY:
Inclusion Criteria:

Caregivers of children who are aged 0-23 months whose eligible child/children slept in the household the night before the survey will be interviewed

Exclusion Criteria:

Caregivers of children who are aged above 23 months

Ages: 0 Days to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100000 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-10-04 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
proportion of identified stakeholders routinely engaged during implementation | 3 months
  Number of identified stakeholders mapped out from inception divided by the Number of identified stakeholders engaged on a routine basis during implementation
Proportion of planned stakeholders engagement meetings conducted | 3 months
  Number of Planned stakeholders engagement meetings planned divided by the Number of planned engagement meetings conducted
Number of households enrolled and receiving DSI's | 6 months
  Number of households successfully enrolled and benefitting from DSI's
Proportions of Health facilities in intervention communities with updated microplans developed with the communities | 3 months
  Number of Health facilities in intervention communities with an updated micro plan co-developed with the participation of the host divided by the Total number of health facilities within the Intervention communities
Proportion of Health facilities in intervention areas conducting vaccination sessions for all catchment areas | 3 months
  Number of Health facilities in intervention areas conducting vaccination sessions for all catchment areas divided by the Total number of Health facilities in intervention Communities implementing DSI's

SECONDARY OUTCOMES:
Cost per individual for enrolment and provision of DSI's | 6-12 months
  Total amount spent on provision of DSI's per country divided by the Total number of individuals provided with DSI's per country
Cost per percentage point increase in coverage | 6-12 months
  Total amount spent on enrolment and Provision of DSI's per cluster divided by percentage increase in coverage per cluster
Proportion of household receiving DSI who feel more accepting of vaccines | 3 months
  Number of households receiving DSI who feel more accepting of vaccines divided by Number of households successfully enrolled and receiving DSI's
Proportion of Households in intervention communities who identify non-cash DSI as a source of Vaccine information | 3 months
  Number of households in intervention communities who identify non-cash DSI as a source of vaccine information divided by the Total number of households surveyed in intervention communities
Proportion of households in intervention communities identifying lack of knowledge as a reason for under-immunization or zero dose | 3 months
  Number of households in intervention communities identifying lack of Knowledge as a reason for under-immunization or zero dose divided by the Total number of households surveyed in intervention communities with under-immunized or Zero dose children
Number of households in intervention communities identifying lack of trust as a reason for under-immunization or zero dose | 3 months
  Number of households in intervention communities identifying lack of trust as a reason for under-immunization or zero dose divided by the Total number of households surveyed in intervention communities with under-immunization or zero dose
Proportion of households in intervention communities identifying lack of motivation as a reason for under-immunization or zero dose | 3 months
  Number of households identifying lack of motivation as a reason for under-immunization or zero dose divided by the Total number of households in intervention communities with under-immunized or zero dose children
Proportion of households in intervention communities with children receiving Vaccines appropriately/timely | 3 months
  Number of households surveyed in intervention communities with eligible children who have been appropriately vaccinated divided by Total Number of households surveyed in intervention communities with eligible children
DTP1 Coverage in Intervention Districts | 3 months
  Number of Children receiving DTP1 vaccinations in intervention districts divided by Total number of eligible children in the intervention districts
DTP3 coverage in intervention districts | 3 months
  Number of Children receiving DTP3 vaccinations in intervention districts divided by Total number of eligible children in the intervention districts
DTP1-DTP3 drop out rate in intervention districts | 3 months
  Difference in the coverage of DTP1 and DTP3 vaccines in intervention districts divided by DTP1 coverage in intervention districts

CONTACTS AND LOCATIONS:
Overall Officials: Obinna Ebirim, MSc, Study Director — Corona Management Systems; Chijioke Kaduru, MPH, Principal Investigator — Corona Management Systems
Locations (2):
- Nigeria (2):
  - Kwara State Prmary Healthcare Development Agency, Ilorin, Kwara State
  - Oyo State Primary Healthcare Board, Ibadan, Oyo State

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahachi K, Kessels J, Boateng K, Jean Baptiste AE, Mitula P, Ekeman E, Nic Lochlainn L, Rosewell A, Sodha SV, Abela-Ridder B, Gabrielli AF. Zero- or missed-dose children in Nigeria: Contributing factors and interventions to overcome immunization service delivery challenges. Vaccine. 2022 Sep 2;40(37):5433-5444. doi: 10.1016/j.vaccine.2022.07.058. Epub 2022 Aug 13. PMID 35973864
- [Background] Equity Reference Group. 2023. ERG Advocacy Brief. Accessed March 06, 2023. https://drive.google.com/file/d/1VpuVX85RWd_vq6FJ4lcmCnPOYJp1AhuM/view
- [Background] District Health Information Systems version 2 (DHIS 2). Federal Ministry of Health. 2023
- [Background] Diphtheria tetanus toxoid and pertussis (DTP) vaccination coverage; https://immunisationdata.who.int/pages/coverage/DTP.html?CODE=NGA&ANTIGEN=DTPCV1&YEAR
- [Background] 2021 Multiple Indicator Cluster Survey (Mics) & National Immunisation Coverage Survey (NICS): Survey Findings Report https://www.unicef.org/nigeria/media/6316/file/2021%20MICS%20full%20report%20.pdf 2022 Aug
- [Background] MOMENTUM. (2021). MOMENTUM Nigeria Country Profile - Immunisation - JSI. https://www.jsi.com/resource/nigeria-country-profile-immunisation/
- [Background] MEDIA FACTSHEET: Takeaways from the 2022 WUENIC estimates for 57 lower-income countries supported by Gavi https://www.gavi.org/news/media-room/media-factsheet-takeaways-2022-wuenic-estimates-57-lower-income-countries-supported
- [Background] United Nations (2022), COVID-19 fuels slowest rate of childhood vaccination in three decades, leaving millions at risk, Health https://news.un.org/en/story/2022/07/1122592
- [Background] UNICEF (2022), Immunisation https://data.unicef.org/topic/child-health/immunisation/
- [Background] WHO (2022), Progress and challenges with Achieving Universal Immunisation Coverage https://www.who.int/publications/m/item/progress-and-challenges